CLINICAL TRIAL: NCT01878812
Title: Immunogenicity and Safety Study of GSK Biologicals' Quadrivalent Split Virion Influenza Vaccine (GSK2321138A) Fluarix/Influsplit Tetra® (2013/2014 Season) in Adults 18 Years of Age and Older
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Quadrivalent Influenza Vaccine, Fluarix/Influsplit Tetra® (2013/2014 Season), in Adults 18 Years of Age and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200188; 2013-001094-25 (EudraCT Number)
Record Dates: First submitted 2013-06-13; First posted 2013-06-17 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-06

CONDITIONS: Influenza
Keywords: Immunogenicity; Influenza; Adults; Safety; Elderly
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

ARMS (2):
- Fluarix/Influsplit Tetra® Adult Group (Experimental): Subjects 18-60 years of age receiving Fluarix/Influsplit Tetra® 2013-2014, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix/Influsplit Tetra® (2013-2014 season)
- Fluarix/Influsplit Tetra® Elderly Group (Experimental): Subjects >60 years of age receiving Fluarix/Influsplit Tetra® 2013-2014, administered intramuscularly in the deltoid region of the non-dominant arm.
  Interventions: Biological: Fluarix/Influsplit Tetra® (2013-2014 season)

INTERVENTIONS:
Biological: Fluarix/Influsplit Tetra® (2013-2014 season) — 1 dose administered intramuscularly in the deltoid region of non-dominant arm

SUMMARY:
The purpose of this study is to assess, in adults 18 years of age and above, the immunogenicity and reactogenicity of the seasonal influenza vaccine, Fluarix/Influsplit Tetra containing the four influenza strains (two A strains and two B strains) for the 2013/2014 season.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* A male or female aged 18 years or above at the time of vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects or subjects with well-controlled chronic diseases as established by medical history and clinical examination before entering the study.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of vaccination.

Exclusion Criteria:

* Participation in previous year's Fluarix registration study (116663).
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within the six months prior to vaccination. Inhaled and topical steroids are allowed.
* Any administration of a long-acting immune-modifying drug within 6 months before study start, or planned administration during the study period.
* Administration of immunoglobulins and/or any blood products within the three months preceding the administration of the study vaccine or planned administration during the study period.
* Administration of an influenza vaccine within the twelve months preceding the study vaccination.
* Receipt of a vaccine other than the study vaccine within 30 days before study vaccination and/or plan to receive any vaccine other than the study vaccine during the entire study period.
* Clinically or virologically confirmed influenza infection within the six months preceding the study vaccination.
* Acute disease and/or fever at the time of enrollment.

  * Fever is defined as temperature ≥ 37.5°C/99.5°F on oral, axillary or tympanic setting, or ≥ 38.0°C/100.4°F on rectal setting. The preferred route for recording temperature in this study will be axillary.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Acute, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Chronic underlying disease (such as cancer, chronic obstructive pulmonary disease under oxygen therapy, insulin-dependent diabetes mellitus), not stabilized or clinically serious.
* History of chronic alcohol consumption and/or drug abuse.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of Guillain-Barré syndrome.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine including latex.
* Anaphylaxis following the administration of vaccine(s).
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study or would make intramuscular injection unsafe.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-07-11 (Actual); Primary Completion 2013-08-05 (Actual); Study Completion 2013-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Started | 60 | 57
Completed | 60 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group | Total
Number analyzed (Participants) | 60 | 57 | 117
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.7 (12.24) | 70.6 (6.81) | 54.24 (18.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Anti-HI Antibody Titers Against 4 Strains of Influenza Disease
Description: The strains assessed were: Flu A/Christchurch/16/2010 H1N1 HI, Flu A/Texas/50/2012 H3N2 HI, Flu B/Massachusetts/2/2012 Yamagata HI, (referred to as Flu B/Mass/2/2012 Yamagata) ,Flu B/Brisbane/60/2008 Victoria HI. Titers are presented as geometric mean titers (GMTs).
Time Frame: At Days 0 and 21
Population: The analysis was based on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects with results available at the specified timepoint.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 60 | 56
Titers
  Flu A/Christchurch/16/2010 H1N1, Day 0 [N=60,56] | 29.8 [20.7 to 42.8] | 14.9 [10.9 to 20.4]
  Flu A/Texas/50/2012 H3N2, Day 0 [N=60,56] | 13.1 [10.1 to 17.0] | 13.5 [10.1 to 18.1]
  Flu B/Mass/2/2012 Yamagata, Day 0 [N=60,56] | 151.0 [111.3 to 204.7] | 110.4 [88.5 to 137.6]
  Flu B/Brisbane/60/2008 Victoria, Day 0 [N=60,56] | 58.5 [44.4 to 77.1] | 56.6 [44.6 to 71.7]
  Flu A/Christchurch/16/2010 H1N1, Day 21 [N=60,56] | 505.0 [400.1 to 637.4] | 230.3 [160.7 to 330.2]
  Flu A/Texas/50/2012 H3N2, Day 21 [N=60,56] | 94.0 [74.1 to 119.3] | 77.9 [58.5 to 103.9]
  Flu B/Mass/2/2012 Yamagata, Day 21 [N=60,56] | 792.6 [661.6 to 949.5] | 535.0 [442.2 to 647.2]
  Flu B/Brisbane/60/2008 Victoria, Day 21 [N=60,56] | 346.9 [288.0 to 417.9] | 239.2 [193.3 to 296.0]

2. Primary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Disease
Description: The strains are: Flu A/Christchurch/16/2010 H1N1 HI, Flu A/Texas/50/2012 H3N2 HI, Flu B/Massachusetts/2/2012 Yamagata HI,(referred to as Flu B/Mass/2/2012 Yamagata), Flu B/Brisbane/60/2008 Victoria HI. A seroprotected subject is defined as a subject with serum HI titre ≥ 1:40.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 60 | 56
Subjects
  Flu A/Christchurch/16/2010 H1N1, Day 0 [N=60,56] | 29 | 12
  Flu A/Christchurch/16/2010 H1N1, Day 21 [N=60,56] | 60 | 49
  Flu A/Texas/50/2012 H3N2, Day 0 [N=60,56] | 12 | 15
  Flu A/Texas/50/2012 H3N2, Day 21 [N=60,56] | 54 | 40
  Flu B/Mass/2/2012 Yamagata, Day 0 [N=60,56] | 56 | 52
  Flu B/Mass/2/2012 Yamagata, Day 21 [N=60,56] | 60 | 56
  Flu B/Brisbane/60/2008 Victoria, Day 0 [N=60,56] | 43 | 40
  Flu B/Brisbane/60/2008 Victoria, Day 21 [N=60,56] | 60 | 55

3. Primary Outcome: Number of Seroconverted Subjects Against 4 Strains of Influenza Disease
Description: The strains are: Flu A/Christchurch/16/2010 H1N1 HI,(referred to as Flu A/Christch/16/2010 H1N1), Flu A/Texas/50/2012 H3N2 HI, Flu B/Massachusetts/2/2012 Yamagata HI, (referred to as Flu B/Mass/2/2012 Yamagata), Flu B/Brisbane/60/2008 Victoria HI. A seroconverted subject is defined as a subject with either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least 4-fold increase in post-vaccination titer.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 60 | 56
Subjects
  Flu A/Christch/16/2010 H1N1, Day 21 [N=60,56] | 48 | 43
  Flu A/Texas/50/2012 H3N2, Day 21 [N=60,56] | 41 | 27
  Flu B/Mass/2/2012 Yamagata, Day 21 [N=60,56] | 35 | 32
  Flu B/Brisbane/60/2008 Victoria, Day 21 [N=60,56] | 37 | 24

4. Primary Outcome: Mean Geometric Increase (MGI) for HI Antibody Titer Against the 4 Flu Strains of Influenza Disease
Description: The strains are: Flu A/Christchurch/16/2010 H1N1 HI, (referred to as Flu A/Christch/16/2010 H1N1), Flu A/Texas/50/2012 H3N2 HI, Flu B/Massachusetts/2/2012 Yamagata HI, (referred to as Flu B/Mass/2/2012 Yamagata) Flu B/Brisbane/60/2008 Victoria HI. MGI was defined as the fold increase in serum HI geometric mean titers post-vaccination compared to Day 0.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 60 | 56
Fold increase
  Flu A/Christch/16/2010 H1N1, Day 21 [N=60,56] | 17.0 [11.6 to 24.8] | 15.4 [10.5 to 22.6]
  Flu A/Texas/50/2012 H3N2, Day 21 [N=60,56] | 7.2 [5.5 to 9.3] | 5.8 [4.3 to 7.8]
  Flu B/Mass/2/2012 Yamagata, Day 21 [N=60,56] | 5.3 [3.8 to 7.2] | 4.8 [3.9 to 6.1]
  Flu B/Brisbane/60/2008 Victoria, Day 21 [N=60,56] | 5.9 [4.4 to 7.9] | 4.2 [3.2 to 5.7]

5. Primary Outcome: Seroprotection Powers (SPP) for HI Antibody Titer Against the 4 Flu Strains of Influenza Disease
Description: The strains are: Flu A/Christchurch/16/2010 H1N1 HI, (referred to as Flu A/Christch/16/2010 H1N1), Flu A/Texas/50/2012 H3N2 HI, Flu B/Massachusetts/2/2012 Yamagata HI, (referred to as Flu B/Mass/2/2012 Yamagata), Flu B/Brisbane/60/2008 Victoria HI. SPP is defined as the percentage of subjects who had a pre-vaccination titer < 1:40 and a post-vaccination titer ≥ 1:40.
Time Frame: During a 4-day follow-up period after vaccination (i.e. day of vaccination and 3 subsequent days)
Population: as for outcome 1
Measure: Number; unit: Percentage of subjects
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 48 | 44
Percentage of subjects
  Flu A/Christch/16/2010 H1N1, Day 21 [N=31,44] | 100 | 84.1
  Flu A/Texas/50/2012 H3N2, Day 21 [N=48,41] | 87.5 | 61.0
  Flu B/Mass/2/2012 Yamagata, Day 21 [N=17, 16] | 100 | 93.8
  Flu B/Brisbane/60/2008 Victoria, Day 21 [N=4,4] | 100 | 100

6. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were ecchymosis, induration, pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 ecchymosis/induration/redness/swelling = ecchymosis/induration/redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During a 21-day follow-up period after vaccination (i.e. day of vaccination and 20 subsequent days)
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 60 | 57
Subjects
  Any Ecchymosis | 0 | 0
  Grade 3 Ecchymosis | 0 | 0
  Any Induration | 6 | 5
  Grade 3 Induration | 0 | 0
  Any Pain | 37 | 19
  Grade 3 Pain | 1 | 0
  Any Redness | 3 | 6
  Grade 3 Redness | 0 | 0
  Any Swelling | 3 | 2
  Grade 3 Swelling | 0 | 0

7. Secondary Outcome: Number of Days of Solicited Local Symptoms
Description: Assessed solicited local symptoms were ecchymosis, induration, pain, redness and swelling. The number of days is expressed as a mean value.
Time Frame: During the entire study period (Days 0 to 21)
Population: The analysis was based on the Total Vaccinated cohort, which included all subjects with the study vaccine administered with the respective symptoms reported.
Measure: Mean (Inter-Quartile Range); unit: Days
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 37 | 19
Days
  Induration [N=6;5] | 1.8 [1.0 to 2.0] | 2.2 [2.0 to 3.0]
  Pain [N=37;19] | 2.2 [2.0 to 3.0] | 1.9 [1.0 to 2.0]
  Redness [N=3;6] | 2.0 [1.0 to 3.0] | 1.5 [1.0 to 2.0]
  Swelling [N=3;2] | 2.7 [2.0 to 3.0] | 2.0 [2.0 to 2.0]

8. Secondary Outcome: Number of Subjects With Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, shivering, sweating and temperature [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)],. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During a 4-day follow-up period after vaccination (i.e. day of vaccination and 3 subsequent days)
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 60 | 57
Subjects
  Any Arthralgia | 3 | 6
  Grade 3 Arthralgia | 1 | 0
  Related Arthralgia | 1 | 4
  Any Fatigue | 10 | 4
  Grade 3 Fatigue | 1 | 0
  Related Fatigue | 8 | 2
  Any Gastrointestinal symptoms | 3 | 2
  Grade 3 Gastrointestinal symptoms | 0 | 0
  Related Gastrointestinal symptoms | 0 | 1
  Any Headache | 9 | 5
  Grade 3 Headache | 1 | 0
  Related Headache | 4 | 4
  Any Myalgia | 14 | 7
  Grade 3 Myalgia | 1 | 0
  Related Myalgia | 12 | 5
  Any Sweating | 2 | 0
  Grade 3 Sweating | 1 | 0
  Related Sweating | 1 | 0
  Any Shivering | 3 | 2
  Grade 3 Shivering | 1 | 0
  Related Shivering | 3 | 2
  Any Temperature | 0 | 0
  Grade 3 Temperature | 0 | 0
  Related Temperature | 0 | 0

9. Secondary Outcome: Number of Days of Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, gastrointestinal symptoms, headache, myalgia, shivering, sweating and temperature [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)],. Any = occurrence of the symptom regardless of intensity grade. The number of days is expressed as a mean value.
Time Frame: During a 4-day follow-up period after vaccination (i.e. day of vaccination and 3 subsequent days)
Population: as for outcome 7
Measure: Mean (Inter-Quartile Range); unit: Days
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 14 | 7
Days
  Arthralgia [N=3;6] | 2.7 [2.0 to 3.0] | 1.8 [1.0 to 2.0]
  Fatigue [N=10;4] | 1.6 [1.0 to 2.0] | 2.8 [2.0 to 3.5]
  Gastrointestinal symptoms [N=3;2] | 2.0 [1.0 to 3.0] | 2.5 [1.0 to 4.0]
  Headache [N=9;5] | 1.9 [1.0 to 2.0] | 1.4 [1.0 to 2.0]
  Myalgia [N=14;7] | 1.8 [1.0 to 2.0] | 2.0 [1.0 to 2.0]
  Sweating [N=3;2] | 1.7 [1.0 to 3.0] | 2.0 [2.0 to 2.0]
  Shivering [N=2;0] | 2.0 [1.0 to 3.0] | NA [NA to NA] — Duration of this symptom was not assessed or confirmation was missing because the symptom was not reported in this group.

10. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During a 4-day follow-up period after vaccination (i.e. day of vaccination and 3 subsequent days)
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 60 | 57
Subjects
  Subjects with any AE(s) | 6 | 9
  Subjects with grade 3 AE(s) | 1 | 0
  Subjects with related AE(s) | 0 | 0

11. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Serious Adverse Events (SAEs).
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: At Days 0 and 21
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 60 | 57
Subjects
  Subjects with any SAE(s) | 0 | 0
  Subjects with related SAE(s) | 0 | 0

12. Secondary Outcome: Anti-HI Antibody Titers Against 4 Strains of Influenza Virus by Vaccination Status
Description: The strains are: Flu A/Christchurch/16/2010 H1N1 HI, (referred to as Flu A/Christch/16/2010 H1N1), Flu A/Texas/50/2012 H3N2 HI, Flu B/Massachusetts/2/2012 Yamagata HI, (referred to as Flu B/Mass/2/2012 Yamagata), Flu B/Brisbane/60/2008 Victoria HI. Titers are presented as geometric mean titers (GMTs). Vaccination status is presented as Y = vaccinated or N = not vaccinated during the 2012-2013 season.
Time Frame: At Days 0 and 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 60 | 56
Titers
  Flu A/Christch/16/2010 H1N1, Day 0,Y [N=12,24] | 65.4 [31.9 to 134.1] | 16.1 [10.5 to 24.7]
  Flu A/Christch/16/2010 H1N1, Day 0,N [N=48,32] | 24.5 [16.2 to 36.8] | 14.1 [8.9 to 22.4]
  Flu A/Texas/50/2012 H3N2, Day 0, Y [N=12.24] | 21.8 [9.5 to 50.0] | 15.0 [9.4 to 23.8]
  Flu A/Texas/50/2012 H3N2, Day 0, N [N=48,32] | 11.5 [8.9 to 15.0] | 12.6 [8.5 to 18.6]
  Flu B/Mass/2/2012 Yamagata, Day 0,Y [N=12,24] | 174.4 [88.4 to 343.8] | 111.6 [83.7 to 148.7]
  Flu B/Mass/2/2012 Yamagata, Day 0,N [N=48,32] | 145.6 [102.4 to 207.1] | 109.5 [78.4 to 152.8]
  Flu B/Brisbane/60/2008 Victoria, Day 0,Y [N=12,24] | 113.2 [67.2 to 190.8] | 62.7 [44.5 to 88.2]
  Flu B/Brisbane/60/2008 Victoria, Day 0,N [N=48,32] | 49.6 [36.4 to 67.6] | 52.4 [37.2 to 73.6]
  Flu A/Christch/16/2010 H1N1, Day 21,Y [N=12,24] | 570.2 [362.2 to 897.4] | 198.6 [111.2 to 355.0]
  Flu A/Christch/16/2010 H1N1, Day 21,N [N=48,32] | 489.9 [372.2 to 644.9] | 257.4 [159.1 to 416.2]
  Flu A/Texas/50/2012 H3N2, Day 21,Y [N=12,24] | 119.9 [67.8 to 211.9] | 68.2 [44.9 to 103.7]
  Flu A/Texas/50/2012 H3N2, Day 21,N [N=48,32] | 88.5 [67.6 to 115.8] | 86.1 [57.3 to 129.6]
  Flu B/Mass/2/2012 Yamagata, Day 21,Y [N=12,24] | 522.9 [316.8 to 863.0] | 415.2 [305.8 to 563.6]
  Flu B/Mass/2/2012 Yamagata, Day 21,N [N=48,32] | 879.5 [729.8 to 1059.9] | 647.0 [511.9 to 817.8]
  Flu B/Brisbane/60/2008 Victoria,Day 21,Y [N=12,24] | 269.0 [188.1 to 384.8] | 162.2 [117.9 to 223.2]
  Flu B/Brisbane/60/2008 Victoria,Day 21,N [N=48,32] | 369.7 [297.6 to 459.1] | 320.0 [248.3 to 412.5]

13. Secondary Outcome: Number of Seroprotected Subjects Against 4 Strains of Influenza Virus by Vaccination Status
Description: The strains are: Flu A/Christchurch/16/2010 H1N1 HI, (referred to as Flu A/Christch/16/2010 H1N1), Flu A/Texas/50/2012 H3N2 HI, Flu B/Massachusetts/2/2012 Yamagata HI, (referred to as Flu B/Mass/2/2012 Yamagata), Flu B/Brisbane/60/2008 Victoria HI. A seroprotected subject is defined as a subject with serum HI titre ≥ 1:40. Vaccination status is presented as Y = vaccinated or N = not vaccinated during the 2012-2013 season.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 60 | 56
Subjects
  Flu A/Christch/16/2010 H1N1, Day 0,Y [N=12,24] | 9 | 5
  Flu A/Christch/16/2010 H1N1, Day 0,N [N=48,32] | 20 | 7
  Flu A/Texas/50/2012 H3N2, Day 0, Y [N=12.24] | 4 | 7
  Flu A/Texas/50/2012 H3N2, Day 0, N [N=48,32] | 8 | 8
  Flu B/Mass/2/2012 Yamagata, Day 0,Y [N=12,24] | 11 | 23
  Flu B/Mass/2/2012 Yamagata, Day 0,N [N=48,32] | 45 | 29
  Flu B/Brisbane/60/2008 Victoria, Day 0,Y [N=12,24] | 11 | 20
  Flu B/Brisbane/60/2008 Victoria, Day 0,N [N=48,32] | 32 | 20
  Flu A/Christch/16/2010 H1N1, Day 21,Y [N=12,24] | 12 | 21
  Flu A/Christch/16/2010 H1N1, Day 21,N [N=48,32] | 48 | 28
  Flu A/Texas/50/2012 H3N2, Day 21,Y [N=12,24] | 11 | 18
  Flu A/Texas/50/2012 H3N2, Day 21,N [N=48,32] | 43 | 22
  Flu B/Mass/2/2012 Yamagata, Day 21,Y [N=12,24] | 12 | 24
  Flu B/Mass/2/2012 Yamagata, Day 21,N [N=48,32] | 48 | 32
  Flu B/Brisbane/60/2008 Victoria,Day 21,Y [N=12,24] | 12 | 23
  Flu B/Brisbane/60/2008 Victoria,Day 21,N [N=48,32] | 48 | 32

14. Secondary Outcome: Number of Seroconverted Subjects Against 4 Strains of Influenza Virus by Vaccination Status
Description: The strains are: Flu A/Christchurch/16/2010 H1N1 HI, (referred to as Flu A/Christch/16/2010 H1N1), Flu A/Texas/50/2012 H3N2 HI, Flu B/Massachusetts/2/2012 Yamagata HI, (referred to as Flu B/Mass/2/2012 Yamagata), Flu B/Brisbane/60/2008 Victoria HI. A seroconverted subject is defined as a subject with either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least 4-fold increase in post-vaccination titer. Vaccination status is presented as Y = vaccinated or N = not vaccinated during the 2012-2013 season.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 60 | 56
Subjects
  Flu A/Christch/16/2010 H1N1, Day 21,Y [N=12,24] | 8 | 18
  Flu A/Christch/16/2010 H1N1, Day 21,N [N=48,32] | 40 | 25
  Flu A/Texas/50/2012 H3N2, Day 21,Y [N=12,24] | 7 | 10
  Flu A/Texas/50/2012 H3N2, Day 21,N [N=48,32] | 34 | 17
  Flu B/Mass/2/2012 Yamagata, Day 21,Y [N=12,24] | 3 | 10
  Flu B/Mass/2/2012 Yamagata, Day 21,N [N=48,32] | 32 | 22
  Flu B/Brisbane/60/2008 Victoria,Day 21,Y [N=12,24] | 2 | 4
  Flu B/Brisbane/60/2008 Victoria,Day 21,N [N=48,32] | 35 | 20

15. Secondary Outcome: Mean Geometric Increase (MGI) for HI Antibody Titer Against the 4 Flu Strains of Influenza Virus by Vaccination Status
Description: The strains are: Flu A/Christchurch/16/2010 H1N1 HI, (referred to as Flu A/Christch/16/2010 H1N1), Flu A/Texas/50/2012 H3N2 HI, Flu B/Massachusetts/2/2012 Yamagata HI, (referred to as Flu B/Mass/2/2012 Yamagata), Flu B/Brisbane/60/2008 Victoria HI. MGI was defined as the fold increase in serum HI geometric mean titers post-vaccination compared to Day 0. Vaccination status is presented as Y = vaccinated or N = not vaccinated during the 2012-2013 season.
Time Frame: At Day 21
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Number analyzed (Participants) | 60 | 56
Titers
  Flu A/Christch/16/2010 H1N1, Day 21,Y [N=12,24] | 8.7 [3.3 to 23.2] | 12.4 [7.1 to 21.6]
  Flu A/Christch/16/2010 H1N1, Day 21,N [N=48,32] | 20.0 [13.2 to 30.3] | 18.2 [10.6 to 31.4]
  Flu A/Texas/50/2012 H3N2, Day 21,Y [N=12,24] | 5.5 [2.5 to 12.0] | 4.6 [2.9 to 7.2]
  Flu A/Texas/50/2012 H3N2, Day 21,N [N=48,32] | 7.7 [5.8 to 10.1] | 6.9 [4.5 to 10.4]
  Flu B/Mass/2/2012 Yamagata, Day 21,Y [N=12,24] | 3.0 [1.6 to 5.7] | 3.7 [2.7 to 5.2]
  Flu B/Mass/2/2012 Yamagata, Day 21,N [N=48,32] | 6.0 [4.2 to 8.6] | 5.9 [4.4 to 7.9]
  Flu B/Brisbane/60/2008 Victoria,Day 21,Y [N=12,24] | 2.4 [1.6 to 3.6] | 2.6 [1.7 to 3.9]
  Flu B/Brisbane/60/2008 Victoria,Day 21,N [N=48,32] | 7.4 [5.4 to 10.3] | 6.1 [4.2 to 8.9]

ADVERSE EVENTS:
Time Frame: Solicited symptoms: Days 0-4 post-vaccination, unsolicited AEs: days 0-21 post-vaccination, SAEs: the entire study duration (Days 0-21 post-vaccination).
Arm/Group | Fluarix/Influsplit Tetra® Adult Group | Fluarix/Influsplit Tetra® Elderly Group
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/57
Other Adverse Events (participants affected / at risk) | 46/60 | 24/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluarix/Influsplit Tetra® Adult Group (N=60) | Fluarix/Influsplit Tetra® Elderly Group (N=57)
Induration (General disorders) | 6 | 5
Pain (General disorders) | 37 | 19
Redness (General disorders) | 3 | 6
Swelling (General disorders) | 3 | 2
Arthralgia (General disorders) | 3 | 6
Fatigue (General disorders) | 10 | 4
Gastrointestinal symptoms (General disorders) | 3 | 2
Headache (General disorders) | 9 | 5
Myalgia (General disorders) | 14 | 7
Sweating (General disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.